CLINICAL TRIAL: NCT03447184
Title: Will Long-term Endogenous Androgen Priming, Using a Combination of Low Dose HCG and Aromatase Inhibitor in Bologna Criteria Poor Responder Patients Increase Ovarian Reserve Parameters - A Pilot Study
Brief Title: Long-term Endogenous Androgen Priming in Bologna Criteria Poor Responder Patients - A Pilot Study
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CS/BVMD/18/01
Record Dates: First submitted 2018-01-23; First posted 2018-02-27 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Poor Ovarian Response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Follicular fluid Granulosa cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Androgen priming: Eight weeks prior to stimulation for IVF - at the onset of menses, patients will start treatment with a low dose of rhCG (Ovitrelle). At the same time daily treatment with the aromatase inhibitor will commence, concomitantly with GnRHa down-regulation with a depot GnRHa (28days). After 8 weeks, a standard rFSH stimulation with either 300 IU rFSH or 300 IU rFSH+rLH will start. The androgen priming (hCG and aromatase inhibitor) will stop on the first day of stimulation.
  Interventions: Drug: Androgen priming

INTERVENTIONS:
Drug: Androgen priming — Androgen priming: with a low dose of recombinant hCG, aromatase inhibitor, and a depot GnRHa for 8 weeks Stimulation: a standard rFSH stimulation with either 300 IU rFSH or 300 IU (rFSH + rLH) Blood sampling: 6 blood samples to measure FSH, LH, E2, testosterone, and AMH Ultrasound examination: to count all antral follicles, 2-10 mm in each ovary Follicular fluid: to analyze E2, androstenedione, testosterone, progesterone, inhibin B.
  Granulosa cells: to analyze gene expression in cumulus and mural granulosa cells of Luteinising hormone receptor (LHR), 3β-hydroxy-steroid-dehydrogenase (3ßHSD), inhibin-Ba (INHB-A) receptor, androgen and FSH receptor
  Other Names: low dose hCG and aromatase inhibitor priming

SUMMARY:
Until now no scientific clinical evidence exists regarding the possible impact of long term endogenous androgen priming in IVF patients aligned with the Bologna Criteria, in specific the impact of priming on serum parameters correlated with the ovarian reserve, antral follicle count, and the number of retrievable follicles. Thus, this pilot-study will explore a new suggested protocol for the Bologna criteria patient developed from basic physiology, and will if successful result in a subsequent randomized controlled trial in the same subset of patients, enabling a possible paradigm shift in the treatment of poor ovarian response (POR).

DETAILED DESCRIPTION:
A single center study pilot study in 30 IVF Bologna criteria POR patients. All patients fulfilling the ESHRE Bologna criteria will be eligible for inclusion.

Eight weeks prior to stimulation for IVF, patients will start treatment with a low dose of rhCG (Ovitrelle). At the same time daily treatment with the aromatase inhibitor daily will commence, concomitantly with GnRHa down-regulation with a depot GnRHa.

After 8 weeks, stimulation will be performed with a fixed dose of 300 IU rFSH (Gonal F, Merck) for the first 5 days in patients ≤ 34 years of age and 300 IU Pergoveris (Merck) in patients ≥ 35 years of age. The use of hCG and aromatase inhibitor will stop on the first day of stimulation.

Monitoring will be performed according to the standard procedure of the clinic. Patients will receive a bolus of 6.500 IU rhCG (Ovitrelle, Merck) for triggering of final oocyte maturation. Oocyte pick-up and embryo transfer will be performed according to the policy of the clinic. Oocyte pick-up (OPU) and embryo transfer will be performed according to standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 41 years
* BMI < 30 kg/m2
* Ovarian reserve, according to the ESHRE Bologna Criteria measured within two months prior to stimulation start

Bologna criteria: At least two of the following three features present:

* Advanced maternal age (≥40 years) or any other risk factor for POR
* A previous POR (≤3 oocytes with a conventional stimulation protocol)
* An abnormal ovarian reserve test (i.e. antral follicle count < 5-7 follicles or AMH< 0.5 - 1.1 ng/mL)
* Poor responder if - Two previous episodes of POR after maximal stimulation (300 IU)

  * Receiving GnRH-antagonist co-treatment during ovarian stimulation
  * Agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
  * Have given written informed consent with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Chronical medical conditions like Diabetes, Crohns disease, Thyroid disease, Hepatitis B and Sexually Transmitted Diseases Simultaneous participation in an interventional clinical trial.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Bologna poor responders: At least two of the following three features present:
  * Advanced maternal age (≥40 years) or any other risk factor for POR
  * A previous POR (≤3 oocytes with a conventional stimulation protocol)
  * An abnormal ovarian reserve test (i.e. antral follicle count < 5-7 follicles or AMH< 0.5 - 1.1 ng/mL)
  * Poor responder if - Two previous episodes of POR after maximal stimulation (300 IU)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of AMH | 8 weeks after starting androgen priming
  Blood sampling

SECONDARY OUTCOMES:
Number of antral follicles | 8 weeks after starting androgen priming
  Follicles 2-10mm on ultrasound
Serum concentrations of testosterone | Up to 2 weeks after starting FSH stimulation
  Blood sampling
Serum concentrations of hCG | Up to 2 weeks after starting FSH stimulation
  Blood sampling
Serum concentrations of progesterone | Up to 2 weeks after starting FSH stimulation
  Blood sampling
Number of antral follicles | Up to 2 weeks after starting FSH stimulation
  Follicles 2-10 mm on ultrasound
Number of pre-ovulatory follicles | Up to 2 weeks after starting FSH stimulation
  Follicles >/= 14 mm on ultrasound

OTHER OUTCOMES:
Follicular fluid concentration of estradiol | Up to one hour after ovum pick-up
  Aspiration of follicular fluid while doing ovum pick-up
Follicular fluid concentration of androstenedione | Up to one hour after ovum pick-up
  Aspiration of follicular fluid while doing ovum pick-up
Follicular fluid concentration of testosterone | Up to one hour after ovum pick-up
  Aspiration of follicular fluid while doing ovum pick-up
Follicular fluid concentration of progesterone | Up to one hour after ovum pick-up
  Aspiration of follicular fluid while doing ovum pick-up
Follicular fluid concentration of inhibin B | Up to one hour after ovum pick-up
  Aspiration of follicular fluid while doing ovum pick-up
Cumulus and mural Luteinising hormone receptor (LHR) gene expression | Up to one hour after ovum pick-up
  Cumulus and mural granulosa cells from oocyte from the first follicle in each women were isolated immediately after ovum pick-up and snap frozen for analysis of LHR gene expression. qPCR was performed and calculation of the expression level of the gene of interest was carried out according to the comparative method, normalised to glyceraldehyde 3-phosphate dehydrogenase (GAPDH) for relative quantification of gene expression.
Cumulus and mural 3β-hydroxy-steroid-dehydrogenase (3ßHSD) gene expression | Up to one hour after ovum pick-up
  Cumulus and mural granulosa cells from oocyte from the first follicle in each women were isolated immediately after ovum pick-up and snap frozen for analysis of 3ßHSD gene expression. qPCR was performed and calculation of the expression level of the gene of interest was carried out according to the comparative method, normalised to glyceraldehyde 3-phosphate dehydrogenase (GAPDH) for relative quantification of gene expression.
Cumulus and mural inhibin-Ba (INHB-A) receptor gene expression | Up to one hour after ovum pick-up
  Cumulus and mural granulosa cells from oocyte from the first follicle in each women were isolated immediately after ovum pick-up and snap frozen for analysis of INHB-A gene expression. qPCR was performed and calculation of the expression level of the gene of interest was carried out according to the comparative method, normalised to glyceraldehyde 3-phosphate dehydrogenase (GAPDH) for relative quantification of gene expression.
Cumulus and mural androgen receptor gene expression | Up to one hour after ovum pick-up
  Cumulus and mural granulosa cells from oocyte from the first follicle in each women were isolated immediately after ovum pick-up and snap frozen for analysis of androgen receptor gene expression. qPCR was performed and calculation of the expression level of the gene of interest was carried out according to the comparative method, normalised to glyceraldehyde 3-phosphate dehydrogenase (GAPDH) for relative quantification of gene expression.
Cumulus and mural FSH receptor gene expression | Up to one hour after ovum pick-up
  Cumulus and mural granulosa cells from oocyte from the first follicle in each women were isolated immediately after ovum pick-up and snap frozen for analysis of FSH receptor gene expression. qPCR was performed and calculation of the expression level of the gene of interest was carried out according to the comparative method, normalised to glyceraldehyde 3-phosphate dehydrogenase (GAPDH) for relative quantification of gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Lan N Vuong, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vuong TNL, Ho MT, Ha TQ, Jensen MB, Andersen CY, Humaidan P. Effect of GnRHa ovulation trigger dose on follicular fluid characteristics and granulosa cell gene expression profiles. J Assist Reprod Genet. 2017 Apr;34(4):471-478. doi: 10.1007/s10815-017-0891-9. Epub 2017 Feb 14. PMID 28197932